CLINICAL TRIAL: NCT02711813
Title: Study to Assess Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of TAB08 in Patients With Systemic Lupus Erythematosus, Not Adequately Controlled With Current Concomitant Therapy
Brief Title: TAB08 in Patients With Systemic Lupus Erythematosus (SLE), Not Adequately Controlled With Current Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Theramab LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAB08-SLE-01
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — TGN-1412

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo to TAB08
  Interventions: Other: Placebo
- TAB08 Dose 1 (Experimental)
  Interventions: Drug: TAB08
- TAB08 Dose 2 (Experimental)
  Interventions: Drug: TAB08

INTERVENTIONS:
Drug: TAB08 — biologic
  Arms: TAB08 Dose 1; TAB08 Dose 2
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether TAB08 may be beneficial compared to placebo in patients with active Systemic Lupus Erythematosus, not adequately controlled with current concomitant treatment. Secondary purpose is to assess efficacy, safety, pharmacokinetic and pharmacodynamic parameters in this study population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Lupus Erythematosus according to American College of Rheumatology (ACR) criteria (4 of 11)
* Active SLE (SLE Disease Activity Index ≥ 6)
* Skin or joint SLE manifestations

Exclusion Criteria:

* Lupus-nephritis and/or central nervous system affection (neuro-lupus)
* Prohibited treatment
* Pregnant or nursing women
* Concomitant systemic therapy dosage modification (if any) within 4 weeks before randomization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number and proportion of treatment responders per SLE Responder Index (SRI) | 24 weeks
Adverse Events | 24 weeks

SECONDARY OUTCOMES:
Patient-reportet health outcome assessed by Short Form - 36 questionnaire (SF-36) | 24 weeks
Area and severity of SLE skin damage by Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniil Nemenov, M.D., Study Director — Theramab LLC
Locations (1):
- Federal State Budget Institution "Research Institute of Rheumatology of V.A. Nasonova" Russian Academy of Medical Sciences, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069